CLINICAL TRIAL: NCT02373514
Title: Intravenous Paracetamol Versus Intravenous Dexketoprofen in Patients Presented With Dysmenorrhea in Emergency Department
Brief Title: IV Paracetamol Versus IV Dexketoprofen in Dysmenorrhea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Cenker Eken, Associate Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 57051259-020/70177
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Acetaminophen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol (Active Comparator): Intravenous 1 gm paracetamol in 100 ml saline with rapid infusion
  Interventions: Drug: Paracetamol
- Dexketoprofen (Active Comparator): Intravenous 50 mg dexketoprofen in 100 ml saline with rapid infusion
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Paracetamol — 1 gr paracetamol in 100 ml saline with rapid infusion
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Dexketoprofen — 50 mg dexketoprofen in 100 ml saline with rapid infusion
  Other Names: Arveles
  Arms: Dexketoprofen

SUMMARY:
Patients presented with dysmenorrhea composed the study population. One gram paracetamol and 50 mg dexketoprofen in 100 ml saline with a rapid infusion were compared in ceasing dysmenorrhea in emergency department.

DETAILED DESCRIPTION:
Patients over 18 years old who presented with dysmenorrhea composed the study population. Patients received pain killer within the last six hours, physical findings consistent with peritoneal irritation, allergy to the study drugs, renal or liver failure, drug addiction, pregnancy or woman with lactation and denied to give inform consent were the exclusion criteria. The pain of the study patients are measured with visual analogue scale at baseline, 15th and 30th minutes. At the end of the 30 minutes, rescue drug need is also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysmenorrhea
* Patients over 18 years old

Exclusion Criteria:

* denied to give inform consent
* Renal or liver failure
* Allergy to the study drugs
* Receiving pain killer within the last 6 hours.
* Physical examination findings consistent with peritoneal irritation
* Pregnancy or patients with lactation
* Drug addiction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 15 minutes
  Change in visual analogue scale at 15th minutes from baseline
Visual Analogue Scale | 30 minutes
  Change in visual analogue scale at 30th minutes from baseline

SECONDARY OUTCOMES:
Rescue drug need | 30 minutes
Adverse effects | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)